CLINICAL TRIAL: NCT02214784
Title: A Randomised Controlled Double-Blind Clinical Study To Evaluate The Safety And Performance Of Neuromuscular Electrical Stimulation (NMES) With The Neurotech Vital Device For The Treatment Of Stress Urinary Incontinence
Brief Title: Neurotech Vital Device For The Treatment Of Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BMR-11-1002; ISRCTN68358784 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2013-09-04; First posted 2014-08-12 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary Incontinence; SUI; Continence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Neurotech Vital Device (Active Comparator): 50% of 140 patients on a 12 week treatment programme with the device used 5 days out of 7 for 30minutes over 12 weeks.
  Interventions: Device: Active Neurotech Vital
- Modified Neurotech Vital Device (Placebo Comparator): 50% of 140 patients on a 12 week treatment programme with the device used 5 days out of 7 for 30 minutes over 12 weeks.
  Interventions: Device: Modified Neurotech Vital Device

INTERVENTIONS:
Device: Active Neurotech Vital — 12 weeks treatment for 30 minutes per day, 5 days out of 7.
  Arms: Active Neurotech Vital Device
Device: Modified Neurotech Vital Device — 12 weeks treatment for 30 minutes per day for 5 days out of 7.
  Arms: Modified Neurotech Vital Device

SUMMARY:
Stress Urinary Incontinence (SUI) is described as an uncontrolled loss of urine which happens when physical activities such as running, jumping and lifting etc are carried out or when increased pressure to the bladder in everyday life is applied by simply sneezing or coughing.

There are various treatment options available - surgical operations, pelvic floor exercises/muscle training and electrical stimulation. This study aims to prove that using the Neurotech Vital device for 12 weeks can stimulate the pelvic floor muscles to strengthen and tone them and in doing so improving stress urinary incontinence. We are comparing the Neurotech Vital device with an altered Neurotech Vital device that does not give the same stimulation treatment. There is a 50% chance of you receiving the altered device, if you do, you will be offered the non-altered Neurotech vital device after your first 12 week treatment programme. Both devices are identical in looks, but give different stimulations through the skin contact electrodes.

DETAILED DESCRIPTION:
The study involves wearing a device that includes a wired garment around the hip and bottom area for a period of 30 minutes, 5 days out of 7, for 12 weeks. During this treatment, electrical stimulation is passed through skin contact electrodes (large sticky black pads) which causes the pelvic floor to contract and relax, without you having to do anything. This treatment is not painful and is very similar to the workout you would get from relaxing and contracting your pelvic floor muscles yourself, however the device produces a much stronger contraction.

The study is open to females who have failed a 6 week exercise programme and have been diagnosed with Stress Urinary Incontinence. It will take place at hospital uro-gynaecology clinics/continence clinics across the United Kingdom. The study could last up to 16 months.

This study is being carried out to further prove that the Neurotech Vital device is an effective way of treating stress urinary incontinence in female participants.The study will look at the results of a 12 week treatment programme with the Neurotech Vital device compared to the modified Neurotech Vital device. It will compare the following:

1. how much urine is lost in a standard 1 minute stress test carried out at the baseline visit (start of the treatment) right through to visit 5 (end of the treatment - 12 weeks).
2. How much improvement is shown in the quality of life questionnaire (this is measured by ticking questions which have scores attached to them and adding up the total score for the questionnaire). This questionnaire asks questions on quality of life which is affected by stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are female and at least 18 years of age.
* Subjects who have signed informed consent form prior to any study related activity.
* Subjects who have previously failed a 6 week volitional pelvic floor muscle training programme or in the Investigators opinion an equivalent lifestyle and exercise programme.
* Subjects who have been clinically diagnosed with stress urinary incontinence and demonstrate a >4g urine leakage following a standardised 1-minute stress test at 1 hour post-bladder filling protocol (1-hour pad weight test). Stress urinary incontinence is defined as complaint of involuntary leakage on effort or exertion, or on sneezing and coughing' (International Continence Society).
* Subjects who have scored at least 18 out of 27 for the Stress Incontinence Questions and are confirmed as having predominant stress urinary incontinence on the Medical, Epidemiologic and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire completed at the screening assessment.
* Subjects with a Body Mass Index of ≤ 40 kg/m2
* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained.
* Subjects who are able to understand this study and are willing to complete all the study assessments.

Exclusion Criteria:

* Subjects who have an existing medical condition that would compromise their participation in the study.
* Subjects who have a physical condition that would make them unable to perform the study procedures.
* Subjects who have any respiratory condition including a chronic cough or history of same.
* Subjects with a history of an underlying neurological condition.
* Subjects with a history of low back pain involving the spinal nerve root.
* Subjects who are currently taking medication, or have taken medication in the last 4 weeks, for urinary incontinence or that effect urinary output function including anti-cholinergics or anti-histamines or any anti-anxiety medications.
* Subjects with a blood clotting disorder or who are taking anti-coagulant medications.
* Subjects who have previously had any uro-gynaecological related surgery excluding hysterectomy.
* Subjects with a clinical diagnosis of prolapse greater than Stage 2.
* Subjects who are pregnant or could be pregnant.
* Subjects who are less than 6 months post-partum or who are lactating.
* Subjects who have any intra-uterine devices or metal implants in the pelvic area, including hip and lumbar spine.
* Subjects with pelvic pain or fibromyalgia or paravaginal defect.
* Subjects with an active implanted medical device (i.e. pacemaker, pump etc).
* Subjects with a history of heart disease or stroke.
* Subjects with a known cancer.
* Subjects with an injury or disability affecting any part of their body which will be in contact with the garment.
* Subjects who are currently involved in any injury litigation claims.
* Subjects who have participated in a clinical study in the last 3 months or any previous clinical study with Bio-Medical Research Ltd.
* Subjects who have been committed to an institution by virtue of an order issued either by the courts or by an authority.
* Any vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. Examples are members of a group with a hierarchical structure, such as medical, pharmacy, dental and nursing students, subordinate hospital and laboratory personnel, employees of the pharmaceutical and medical device industry, members of the armed forces, and persons kept in detention. Other vulnerable subjects include patients with incurable diseases, persons in nursing homes, unemployed or impoverished persons, patients in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, minors, and those incapable of giving consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
All participants taking part in a standardised 1-minute stress test | 12 weeks
  We will look at the amount of urine in grams which is lost by participants when carrying out a stress test with all participants and compare their urine loss measured at baseline and then what it measures at 12 weeks after the 12 weeks treatment with the device. Comparing these against one another to look at any improvement.
All participants to complete a Quality of life questionnaire (I-QOL) | 12 weeks
  We will look at the scores which are taken from these questionnaires (depending on which answer is ticked by the participant on the questionnaire) at baseline before treatment with the device commences and then again after 12 weeks of treatment with the device and compare the scores for any improvement.

SECONDARY OUTCOMES:
participants taking part in a 1 minute stress test | 4, 8, 12 and 26 weeks
  We will look at the amount of urine in grams which is lost by participants when carrying out a stress test with all participants and compare their urine loss measured at 4, 8 and 12 weeks against each other and calculate any difference to ascertain if any improvment has been gained by following the device treatment schedule.
participants taking part in a 1-hour pad weight test | Stress test done at 4, 8 and 12 weeks during treatment with the device and at 6 months, for the main and cohort part of study
  The loss of urine in grams after this test at the above time points will be collected and using the definition of dryness (pad weight of less than 1 gram) they will be looked at to see if at any of the above timepoints the participants are classed as dry i.e. have urine loss of less than 1gram following the stres test.
particpants taking part in the stress test and then having the pad weight to show loss of urine. | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  We are looking at a significant reduction in the weight of the pad after the stress test has taken place, this improvement is defined as a greater than 50% reduction in pad weight in all particpants who took the test at baseline compared to the weight of the pad at 4, 8 and 12 weeks and at 6months for the main and cohort studies.
1-hour pad weight test | 4, 8 and 12 weeks and at 6 months, for main and cohort part of the study
  reduction in pad weight on the 1-hour pad weight test in relation to the mean intensity of the stimulation delivered during the 12-week treatment programme;
quality of life questionnaire | 4, 8 and 12 weeks and at 6 months, for main part and cohort part of the study
  quality of life assessed using the Incontinence Quality of Life Questionnaire (I-QOL) (except for the 12 week assessment which is one of the primary endpoints);
quality of life questionnaire | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  quality of life questionnaire assessed using the Kings Health Questionnaire (KHQ)
24 hour pad weight test | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  urine leakage experienced by the subject at home during a 24-hour period (24-hour pad weight test);
24 hour pad weight test | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  dryness, defined as a pad weight of less than 1.3g on the 24-hour pad weight test;
24hour pad weight test | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  significant improvement, defined as a greater than 50% reduction in pad weight from baseline on the 24-hour pad weight test;
3-day diary card | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  number of incontinence episodes/day recorded using a 3-day voiding diary;
3-day voiding diary | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  number of pads used/day recorded using a 3-day voiding diary;
Modified Oxford Score | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  pelvic floor strength and quality of contraction measured using the Modified Oxford Score;
Pelvic floor ultrasound | 4, 8 and 12 weeks and at 6 months for main and cohort part of the study
  pelvic floor muscle function measured using sonographic/real time ultrasound imaging/recording with displacement measurement using on screen callipers on the sonogram unit to assess volitional contractions
participants taking part in a 1 minute stress test | We will compare the urine loss against the urine loss after 4weeks treatment with the device and also after 8weeks treatment with the device and 12 weeks treatment
  We will look at the amount of urine in grams which is lost by participants when carrying out a stress test with all participants and compare their urine loss measured at 4, 8 and 12 weeks against each other and calculate any difference to ascertain if any improvment has been gained by following the device treatment schedule.

OTHER OUTCOMES:
3-day voiding diary | 6, 9 and 12 months
  time to achieve dryness (i.e. no record of any leaks) on the 3-day voiding diary;
device compliance download | 6, 9 and 12 months
  compliance with the treatment protocol during the 12-week treatment programme;
Device Ease of Use Questionnaire | 12 weeks cohort and main study
  subject feedback on the device recorded by the Device Ease of Use Questionnaire following completion of the 12-week treatment programme;
We will collect from all participants the number of Adverse Events (AEs), Serious Adverse Events (SAEs), Serious Adverse Device Events (SADEs) and Uunexpected Adverse Device Events (UADE)and any Device Deficiencies. | Screening to 26 weeks
  the safety will be ascertained according to how many participants report any device related adverse events and and device related serious adverse events also we will look at device deficiencies reported by all the participants
Participants completing a Quality of life questionnaire | scores looked at from the questionnaires completed at 9 months and 12 months
  The scores collected on these questionnaires will be compared against the scores collected at 12 months - The Kings Health Questionnaire and Incontinence Quality of Life Questionnaire (I-QOL)both are completed at 9 months into the study and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: R Tunn, Professor, Principal Investigator — St Hedwig Krankenhaus, Berlin
Locations (3):
- Germany (3):
  - St Hedwig Krankenhaus, Berlin
  - Klinikum Brandenburg,, Brandenburg
  - St Joesph Hospital,, Frankfurt